CLINICAL TRIAL: NCT02340819
Title: A 4-Stage, Open-label, Multicenter Study Including Long-term Extension to Evaluate the Safety, Efficacy and Pharmacokinetics of Teduglutide in Japanese Subjects With PN-dependent Short Bowel Syndrome
Brief Title: Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Teduglutide in Japanese Subjects With PN-dependent Short Bowel Syndrome (SBS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED-C14-004
Record Dates: First submitted 2014-11-13; First posted 2015-01-19 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): 0.05 mg/kg/day administered by subcutaneous injection over a 24-week period.
  Interventions: Drug: Teduglutide

INTERVENTIONS:
Drug: Teduglutide — 0.05 mg/kg/day administered by subcutaneous injection over a 24-week period.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of an investigational treatment (teduglutide) in Japanese patients with PN-dependent SBS. This study will also look at how teduglutide moves through the body (pharmacokinetics).

ELIGIBILITY:
This study has 3 stages, consisting of an optimization/stabilization period (Stage 1), a 24-week treatment period in which all patients will receive teduglutide (Stage 2), and a long-term extension (Stage 3).

During the long-term extension (Stage 3), patients will continue to receive teduglutide for up to an additional 24 months or until teduglutide is commercially available, whichever comes earlier.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- Japan (5):
  - Tohoku University Hospital, Sendai, Aoba-ku
  - Yokohama Municipal Citizen's Hospital, Yokohama, Hodogaya-ku
  - Hospital of Hyogo College of Medicine, Hyōgo, Nishinomiya
  - Osaka University Hospital, Department of Gastroenterological Surgery, Osaka, Suita
  - Osaka University Hospital, Department of Pediatric Surgery, Osaka, Suita

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites, …)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at five centers in Japan between 18 December 2014 (first participant first visit) and 12 November 2018 (last participant last visit).
Pre-assignment Details: Screened participants underwent a maximum 8 week parenteral support (PS) optimization period and 4 to 8 week stabilization period (stage 1) followed by 24 weeks treatment period (stage 2), and a long-term extension period were all participants received same treatment of stage 2 in stage 3 and stage 4. Total study duration was up to 47 months.
Groups:
- Teduglutide: Optimized and stabilized participants received subcutaneous (SC) injection of teduglutide at a dose of 0.05 milligram per kilogram per day (mg/kg/day) once daily for 24 weeks during stage 2, an additional 24 months in stage 3 and continued (stage 4) until the participants entered the long-term extension study SHP633-307 (NCT03596164) or discontinued.
Period: Overall Study
Arm/Group | Teduglutide
Started | 11
Started Stage 2 | 11
Completed Stage 2 | 9
Started Stage 3 | 8
Completed Stage 3 | 7
Started Stage 4 | 7
Completed Stage 4 | 7
Completed | 7
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Discontinued with other reason | 1

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all participants in the intent-to-treat (ITT) population who received at least one dose of study drug. ITT population consists of all participants who are enrolled and eligible to enter Stage 2.
Arm/Group | Teduglutide
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.9 (12.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Stage 2: Absolute Change From Baseline in Weekly Parenteral Support (PS) Volume at Week 24
Description: Absolute change from baseline in weekly PS volume at Week 24 was reported.
Time Frame: Baseline (stage 2), Week 24
Population: Intent-to-treat (ITT) population consisted of all participants who were enrolled and eligible to enter Stage 2. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Liter per week (L/week)
Arm/Group | Teduglutide
Number analyzed (Participants) | 9
Liter per week (L/week) | -4.92 (4.749)

2. Primary Outcome: Stage 2: Percent Change From Baseline in Weekly Parenteral Support (PS) Volume at Week 24
Description: Percent change from baseline in weekly PS volume at Week 24 was reported.
Time Frame: Baseline (stage 2), Week 24
Population: ITT population consisted of all participants who were enrolled and eligible to enter Stage 2. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change in PS volume
Arm/Group | Teduglutide
Number analyzed (Participants) | 9
Percent change in PS volume | -30.07 (25.892)

3. Primary Outcome: Stage 2: Percentage of Participants Who Demonstrate Response to Teduglutide at End of Stage 2
Description: Response was defined as the achievement of at least a 20% reduction from baseline (Visit 2) in weekly PS volume at Week 20 and again at Week 24.
Time Frame: End of Stage 2 (up to Week 24)
Population: ITT population consisted of all participants who were enrolled and eligible to enter Stage 2.
Measure: Number; unit: Percentage of Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 11
Percentage of Participants
  PS Response: Yes | 45.5
  PS Response: No | 54.5

4. Primary Outcome: Stage 2: Absolute Change From Baseline in Number of Days Per Week of Parenteral Support (PS) Usage at Week 24
Description: Absolute change from baseline in number of days per Week of PS usage at Week 24 was reported.
Time Frame: Baseline (stage 2), Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days per week (days/week)
Arm/Group | Teduglutide
Number analyzed (Participants) | 9
Days per week (days/week) | -1.0 (1.80)

5. Primary Outcome: Stage 2: Absolute Change From Baseline in Plasma Citrulline Levels at Week 24
Description: Plasma citrulline was measured as an assessment of enterocyte mass. Absolute change from baseline in plasma citrulline levels at Week 24 was reported.
Time Frame: Baseline (stage 2), Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Teduglutide
Number analyzed (Participants) | 9
Micromoles per liter | 15.0 (17.37)

6. Primary Outcome: Stage 2: Percent Change From Baseline in Plasma Citrulline Levels at Week 24
Description: Plasma citrulline was measured as an assessment of enterocyte mass. Percent change from baseline in plasma citrulline at Week 24 was reported.
Time Frame: Baseline (stage 2), Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Teduglutide
Number analyzed (Participants) | 9
Percent change | 86.9 (112.33)

7. Primary Outcome: Stage 2: Number of Participants Who Achieved Enteral Autonomy at Week 24
Description: Enteral autonomy was defined as no prescribed PS and no use of PS recorded in the participant diary at the end of stage 2. Number of participants who achieved enteral autonomy at Week 24 was reported.
Time Frame: Week 24
Population: ITT population consisted of all participants who were enrolled and eligible to enter Stage 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 11
Participants | 0

8. Primary Outcome: Stage 3: Absolute Change From Baseline in Weekly Parenteral Support (PS) Volume at Extension Month 24
Description: Absolute change from baseline in weekly PS volume at extension Month 24 was reported. Extension month 24 = 30 months of teduglutide treatment.
Time Frame: Baseline (stage 3), Extension Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/week
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
L/week | -8.33 (5.940)

9. Primary Outcome: Stage 3: Percent Change From Baseline in Weekly Parenteral Support (PS) Volume at Extension Month 24
Description: Percent change from baseline in weekly PS volume at extension Month 24 was reported. Extension month 24 = 30 months of teduglutide treatment.
Time Frame: Baseline (stage 3), Extension Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change in PS volume
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Percent change in PS volume | -53.53 (33.866)

10. Primary Outcome: Stage 3: Absolute Change From Baseline in Number of Days Per Week of Parenteral Support (PS) Usage at Extension Month 24
Description: Absolute change from baseline in number of days per Week of PS usage at extension Month 24 was reported. Extension month 24 = 30 months of teduglutide treatment.
Time Frame: Baseline (stage 3), Extension Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
days/week | -2.1 (3.34)

11. Primary Outcome: Stage 3: Absolute Change From Baseline in Plasma Citrulline Levels at Extension Month 24
Description: Plasma citrulline was measured as an assessment of enterocyte mass. Absolute change from baseline in plasma citrulline levels at extension Month 24 was reported. Extension month 24 = 30 months of teduglutide treatment.
Time Frame: Baseline (stage 3), Extension Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Micromoles per liter | 28.3 (24.05)

12. Primary Outcome: Stage 3: Percent Change From Baseline in Plasma Citrulline Levels at Extension Month 24
Description: Plasma citrulline was measured as an assessment of enterocyte mass. Percent change from baseline in plasma citrulline at extension Month 24 was reported. Extension month 24 = 30 months of teduglutide treatment.
Time Frame: Baseline (stage 3), Extension Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Percent change | 135.0 (84.17)

13. Primary Outcome: Stage 4: Absolute Change From Baseline in Weekly Parenteral Support (PS) Volume at End of Treatment
Description: Absolute change from baseline in weekly PS volume at end of treatment was reported.
Time Frame: Baseline (stage 4), End of Treatment (up to 47 months)
Population: ITT population consisted of all participants who were enrolled and eligible to enter Stage 2.
Measure: Mean (Standard Deviation); unit: L/week
Arm/Group | Teduglutide
Number analyzed (Participants) | 11
L/week | -5.08 (6.404)

14. Primary Outcome: Stage 4: Percent Change From Baseline in Weekly Parenteral Support (PS) Volume at End of Treatment
Description: Percent change from baseline in weekly PS volume at end of treatment was reported.
Time Frame: Baseline (stage 4), End of Treatment (up to 47 months)
Population: ITT population consisted of all participants who were enrolled and eligible to enter Stage 2.
Measure: Mean (Standard Deviation); unit: Percent change in PS volume
Arm/Group | Teduglutide
Number analyzed (Participants) | 11
Percent change in PS volume | -34.12 (38.877)

15. Primary Outcome: Stage 4: Absolute Change From Baseline in Number of Days Per Week of Parenteral Support (PS) Usage at End of Treatment
Description: Absolute change from baseline in number of days per week of PS usage at end of treatment was reported.
Time Frame: Baseline (stage 4), End of Treatment (up to 47 months)
Population: ITT population consists of all participants who were enrolled and eligible to enter Stage 2.
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Teduglutide
Number analyzed (Participants) | 11
days/week | -1.4 (2.80)

16. Primary Outcome: Stage 4: Absolute Change From Baseline in Plasma Citrulline Levels at End of Treatment
Description: Plasma citrulline was measured as an assessment of enterocyte mass. Absolute change from baseline in plasma citrulline levels at end of treatment was reported.
Time Frame: Baseline (stage 4), End of Treatment (up to 47 months)
Population: ITT population consisted of all participants who were enrolled and eligible to enter Stage 2.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Teduglutide
Number analyzed (Participants) | 11
Micromoles per liter | 19.3 (19.96)

17. Primary Outcome: Stage 4: Percent Change From Baseline in Plasma Citrulline Levels at End of Treatment
Description: Plasma citrulline was measured as an assessment of enterocyte mass. Percent change in plasma citrulline from baseline at end of treatment was reported.
Time Frame: Baseline (stage 4), End of Treatment (up to 47 months)
Population: ITT population consisted of all participants who were enrolled and eligible to enter Stage 2.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Teduglutide
Number analyzed (Participants) | 11
Percent change | 110.3 (98.13)

18. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC0-Inf) of Teduglutide in Plasma
Description: Area under the concentration-time curve from time zero to infinity of teduglutide in plasma were evaluated.
Time Frame: Pre-dose, 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dose
Population: Pharmacokinetic (PK) analysis population was defined as all participants, at Stage 2, in the safety analysis population for whom the primary PK data were considered sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: Nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Teduglutide
Number analyzed (Participants) | 8
Nanogram*hour per milliliter (ng*h/mL) | 204 (51.1)

19. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to the Last Time Point (AUC0-t) of Teduglutide in Plasma
Description: Area under the concentration-time curve from time zero to the last time point of teduglutide in plasma were evaluated.
Time Frame: Pre-dose, 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dose
Population: PK analysis population was defined as all participants, at Stage 2, in the safety analysis population for whom the primary PK data were considered sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Teduglutide
Number analyzed (Participants) | 8
ng*h/mL | 201 (51.6)

20. Secondary Outcome: Maximum Concentration (Cmax) of Teduglutide in Plasma
Description: Maximum concentration of teduglutide in plasma were evaluated.
Time Frame: Pre-dose, 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Teduglutide
Number analyzed (Participants) | 8
Nanogram per milliliter (ng/mL) | 49.7 (19.7)

21. Secondary Outcome: Time to Reach Maximum Observed Drug Concentration (Tmax) of Teduglutide in Plasma
Description: Time to reach maximum observed drug concentration of teduglutide in plasma was evaluated.
Time Frame: Pre-dose, 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dose
Population: as for outcome 19
Measure: Median (Full Range); unit: hour
Arm/Group | Teduglutide
Number analyzed (Participants) | 8
hour | 2.49 [1.17 to 4.00]

22. Secondary Outcome: Terminal Half-Life (t1/2) of Teduglutide in Plasma
Description: Terminal half-life of teduglutide in plasma were evaluated.
Time Frame: Pre-dose, 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dose
Population: as for outcome 19
Measure: Median (Full Range); unit: hour
Arm/Group | Teduglutide
Number analyzed (Participants) | 8
hour | 1.06 [0.62 to 2.63]

23. Secondary Outcome: Apparent Clearance (CL/F) of Teduglutide in Plasma
Description: Apparent clearance of teduglutide in plasma were evaluated.
Time Frame: Pre-dose, 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dose
Population: PK analysis population was defined as all participants, at Stage 2, in the safety analysis population for whom the primary PK data are considered sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Arm/Group | Teduglutide
Number analyzed (Participants) | 8
liter per hour (L/h) | 14.5 (4.09)

24. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Teduglutide in Plasma
Description: Apparent volume of distribution of teduglutide in plasma were evaluated.
Time Frame: Pre-dose, 15, 30, 60 minutes, 2, 3, 4, 6, 8, 10 and 12 hours post-dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Teduglutide
Number analyzed (Participants) | 8
liter | 27.8 (22.5)

ADVERSE EVENTS:
Time Frame: From start of study treatment up to end of the study (up to 47 months)
Arm/Group | Teduglutide
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 7/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teduglutide (N=11)
Thrombophlebitis (Vascular disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Device occlusion (General disorders) | 1 (2)
Pyrexia (General disorders) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 7 (19)
Sepsis (Infections and infestations) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teduglutide (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vascular pain (Vascular disorders) | 2 (3)
Thyroid cyst (Endocrine disorders) | 1 (1)
Asthenopia (Eye disorders) | 1 (2)
Dry eye (Eye disorders) | 1 (1)
Eye oedema (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Vitreous opacities (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (2)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (7)
Pancreatic duct dilatation (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Toothache (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)
Catheter site inflammation (General disorders) | 1 (1)
Catheter site pain (General disorders) | 2 (3)
Chest pain (General disorders) | 1 (1)
Device occlusion (General disorders) | 3 (4)
Fatigue (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Injection site reaction (General disorders) | 2 (2)
Injury associated with device (General disorders) | 1 (1)
Malaise (General disorders) | 1 (2)
Oedema (General disorders) | 1 (1)
Puncture site pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (7)
Thirst (General disorders) | 1 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Balanitis candida (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 2 (3)
Gingivitis (Infections and infestations) | 1 (2)
Influenza (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (15)
Oral candidiasis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Trichophytosis (Infections and infestations) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Stoma site reaction (Injury, poisoning and procedural complications) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Carcinoembryonic antigen increased (Investigations) | 1 (1)
Intestinal transit time increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Urine output decreased (Investigations) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypozincaemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Dyslalia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (10)
Presyncope (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2)
Anxiety disorder (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT02340819/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT02340819/SAP_001.pdf